CLINICAL TRIAL: NCT04595097
Title: Adjunctive Inspiratory Muscle Training for Patients With COVID-19
Brief Title: Inspiratory Muscle Training in COVID-19 Patients
Acronym: ADDIMTCOVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Ciencias da Saude (Other)
Collaborators: University of Brasilia (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Vinicius Zacarias Maldaner da silva, PhD, Escola Superior de Ciencias da Saude
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CNPQ092020
Record Dates: First submitted 2020-10-19; First posted 2020-10-20 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Covid19; Exercise
Keywords: respiratory function tests; inspiratory muscle training
MeSH Terms: conditions — COVID-19; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The training volume will be 24 sessions. Training frequency will be 3 sessions per week. Duration of training sessions will be around 60min. Patients will perform endurance training or interval training at moderate to high intensities. IMT in both groups will be performed using the PowerBreathe KHP2 device (POWERbreatheKHP2, HaB, International, Southam, UK). Training intensity in the intervention group will be set initially at a load of 50% of patients' maximal inspiratory mouth pressure (MIP). This initial load will be continuously and gradually increased to the highest tolerable intensity during each of the supervised sessions.
  Interventions: Device: inspiratory muscle traiing
- Control group (Active Comparator): The training volume will be 24 sessions. Training frequency will be 3 sessions per week. Duration of training sessions will be around 60min. Patients will perform endurance training or interval training at moderate to high intensities. Sham IMT will be performed using the PowerBreathe KHP2 device (POWERbreatheKHP2, HaB, International, Southam, UK). Training intensity in the control group will be set at 10% baseline PImax and will be not modified throughout the intervention period.
  Interventions: Device: inspiratory muscle traiing

INTERVENTIONS:
Device: inspiratory muscle traiing — The patients are encouraged to inhale against a load to increase the inspiratory muscle strength and endurance
  Other Names: tapered flow resistive loading

SUMMARY:
This study aims to investigate whether adjunctive inspiratory muscle training (IMT) can enhance the benefits of pulmonary rehabilitation (PR) in patients with COVID-19. 120 patients will be randomized into an interventional group (PR plus IMT) and a control group (sham IMT plus PR). Improvement in quality of life, peak VO2 and VE/VCO2 slope will be defined as a primary outcome. Maximal inspiratory pressure, inspiratory muscle endurance, pulmonary function testing, severity of fatigue, cost-effectiveness and six minute walk test will be defined as the secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

To be eligible, participants must be:

* over 18 years of age
* confirmed COVID-19 diagnosis
* Individuals that required hospitalization and either i) non-invasive respiratory support (CPAP, high-flow oxygen catheter, non-breathing oxygen mask, or ii) invasive mechanical ventilation within three months of study recruitment.

Exclusion Criteria:

* Pregnancy
* Dependence on others to perform activities of daily living during the month prior to the current ICU admission (gait aids are acceptable)
* documented cognitive impairment
* Proven or suspected spinal cord injury, or other neuromuscular diseases that will result in a permanent or prolonged weakness (not including ICU acquired weakness)
* Severe neurological disease
* Death is deemed inevitable as a result of the current illness and either the patient or treating clinical or substitute decision-maker are not committed to full active treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary Exercise Testing Measurements | change from baseline in Peak VO2, VE/VCO2 slope and VAT at 8 weeks and 6 months
  Peak VO2 is a measurement of oxygen consumption rate during exercise (milliliters of oxygen per minute). It is calculated by continuous measurement of oxygen consumed during exercise while patients breath through a mask/tube. To account for variability in patient size, the oxygen consumption is divided by patient body weight.The VE/VCO2 slope is calculated as the ratio of minute ventilation (VE) and carbon dioxide production (VCO2). Because these measurements share the same units, the resultant ratio is unitless.The ventilatory anaerobic threshold (VAT) will be determined by the V-slope method.

SECONDARY OUTCOMES:
severity of fatigue | change from baseline in FSS score at 8 weeks and 6 months
  Fatigue severity scale (FSS) is a questionnaire consisting of 9 questions showing the degree of fatigue of patients. An average score of less than 2.8 indicates no fatigue, and more than 6.1 indicates chronic fatigue syndrome
Anxiety and Depression | Change from baseline in HADS score at 8 weeks and 6 months
  Hospital anxiety and depression scale (HADS) is a 14-item questionnaire for screening anxiety (7 items) and depression (7 items). Each item is scored from 0-3 (a 4-point severity scale). Highest anxiety or depression score is 21. Patients are defined as having anxiety or depression or both if the score is 8 or more in the each subscale.
incremental cost-utility ratio | 6 months
  Utility will be measured by Quality Adjusted Life Year (QALYs) as estimated from responses to the Euroqol-5 Dimensions (EQ-5D 5L) health-related quality of life questionnaire. The questionnaire focuses on 5 dimensions: mobility, personal autonomy, current activities, pain/discomfort and anxiety/depression. For each of these dimensions, 5 answers are possible.
Health- related quality of life | change from baseline in EQ-5D score at 8 weeks and 6 months
  EQ-5D is a standardized tool for the assessment of quality of life in 5 different dimensions (Mobility, Self-Care, Usual Activities, Pain/Discomfort, Anxiety/Depression). Possible scores range from 1 (No problem) to 3 (Extreme problems) and each dimension are evaluated individually
Pulmonary function testing | change from baseline in FEV1 and FVC in Liters at 8 weeks and 6 months.
  Spirometry will be performed with a spirometer (Microlab 3.500; CareFusion, Yorba Linda, CA, USA). Three forced expiration maneuvers will be performed for validity and reproducibility purposes according to ATS/ERS criteria, with patients sitting, in a room with controlled temperature, ambient pressure, and relative humidity. The following variables will be analyzed: (a) forced vital capacity (FVC, L), (b) forced expiratory volume in the first second (FEV1, L).
Dyspnea | change from baseline in mMRC score at 8 weeks and 6 months
  The modified Medical Research Council Dyspnea Scale (mMRC). A score from 0-4 is used to classify the impact of dyspnea on physical function in patients with respiratory limitations. 0 represents a person who suffers from dyspnea only with strenuous exercise. 4 represents a person who are to breathless to leave the house, or breathless when dressing/undressing.
Respiratory muscle strength | change from baseline in MIP and MEP at 8 weeks and 6 months
  Pulmonary function test with Maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) measurements
Postural Control | change from baseline in Postural stability test and fall risk test at 8 weeks
  postural control assessed by stabilometry test
isometric knee extension strength | change from baseline in Nm at 8 weeks
  peripheral muscle stregnth assessed by isometric load dynamometer
displacement | change from baseline in CM2 at 8 weeks
  outcomes assessed by baropodometry
trajectory | change from baseline in CM2 at 8 weeks
  outcome assessed by baropodometry
isometric knee flexion strength | change from baseline in Nm at 8 weeks
  peripheral muscle stregnth assessed by isometric load dynamometer
dynamic balance | change from baseline in Total score at 8 weeks
  dynamic balance assessed by Mini-BEST testing
Sit to Stand Test | change from baseline in repetitions at 8 weeks
  exercise capacity assessed by Sit to Stand test

CONTACTS AND LOCATIONS:
Locations (1):
- Secretaria de Saúde do Distrito Federal, Brasília, Federal District, Brazil

REFERENCES:
- [Derived] Maldaner V, Coutinho J, Santana ANDC, Cipriano GFB, Oliveira MC, Carrijo MM, Lino MEM, Cahalin LP, Lima AG, Borges R, Santos DB, Silva IO, Oliveira LVF, Cipriano G Jr. Adjunctive inspiratory muscle training for patients with COVID-19 (COVIDIMT): protocol for randomised controlled double-blind trial. BMJ Open. 2021 Sep 22;11(9):e049545. doi: 10.1136/bmjopen-2021-049545. PMID 34551948